CLINICAL TRIAL: NCT01822548
Title: Randomized, Open Label, Two Parallel Arms, Intervention Trial Comparing the Effect of DPP-IV Inhibitor Vildagliptin vs. Glibenclamide on Circulating Endothelial Progenitor Cell Number in Patients With Type 2 Diabetes in Metformin Failure
Brief Title: Effect of Vildagliptin vs. Glibenclamide on Circulating Endothelial Progenitor Cell Number Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Ivana Zavaroni, Prof., Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-005399-32
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes
Keywords: EPC; diabetes; DPP IV inhibitors
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Vildagliptin; Glyburide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vildagliptin & metformin (Experimental): Vildagliptin 100 mg tablet and metformin (max dose=2500 mg) tablet daily oral administration
  Interventions: Drug: Vildagliptin; Drug: Metformin
- Glibenclamide & metformin (Active Comparator): Glibenclamide maximum dose of 10 mg tablet and metformin (max dose=2500 mg) tablet daily oral administration
  Interventions: Drug: Glibenclamide; Drug: Metformin

INTERVENTIONS:
Drug: Vildagliptin — 100 mg daily
  Other Names: LAF237A
  Arms: Vildagliptin & metformin
Drug: Glibenclamide — 2.5 mg (total daily), progressively increased up to a maximum dose of 5 mg x 2/ day.
  Arms: Glibenclamide & metformin
Drug: Metformin — concomitant therapy with metformin is present in each arm (MAX dose: 2500 mg/die)

SUMMARY:
The purpose of this study is to evaluate the effect of Dipeptidyl peptidase (DPP) -IV inhibitor Vildagliptin vs. Glibenclamide on circulating endothelial progenitor cells (EPCs) number in type 2 diabetes patients in metformin failure. Subjects will be followed for 12 months after randomization.

DETAILED DESCRIPTION:
Diabetic patients show a higher cardiovascular risk compared with non-diabetic patients. It is therefore crucial that blood glucose lowering drugs reveal a favorable cardiovascular risk profile independently of metabolic control.

EPCs are a subset of circulating mononuclear cells derived from the bone marrow. EPCs play a fundamental role in the formation of new blood vessels (neo-endothelization) and repairing of existing blood vessels (re-endothelization) in order to maintain endothelial homeostasis and integrity. Endothelial damage and tissue ischemia, through the release of growth factors and cytokines, represent a strong stimulus for the mobilization of EPCs from the bone marrow. Reduced EPC number has been related to the presence of traditional risk factors for cardiovascular disease and to the development of atherosclerosis and has been shown to predict cardiovascular (CV)risk. Type 2 diabetes is known to be associated with an increased CV risk and a reduced EPC number. Recent data suggest that DPP-IV inhibitors might be involved in the mechanisms promoting bone-marrow EPC mobilization. This putative ancillary effect of DPP-IV might have a favorable impact on type 2 diabetes, a condition characterized by an increased CV risk.

This is a randomized, open-label, active-treatment-controlled, two parallel arm (2:1), intervention trial comparing DPP-IV inhibitor Vildagliptin (100 mg daily) with Glibenclamide (maximum daily dose of 10 mg). Treatment allocation and titration regimens are not blinded.

Primary end-point:Absolute change in the EPC number at visit: V0 (randomization), V2 (month 4), V3 (month 8) and V4 (month 12).

Secondary end-point: Absolute change in HbA1C compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or above 35 years;
* Diagnosis of type 2 diabetes mellitus as defined by the American Diabetes Association , with at least one year of disease duration at the time of the screening visit;
* Blood glucose lowering treatment with Metformin alone (monotherapy) at a stable dose of at least 1.5 g/day (or maximum tolerated dose) in the 3 months prior to the screening visit;
* Insufficient metabolic control as defined by recent (last six months) HbA1c ≥ 7% in any peripheral laboratory and confirmed at the time of the screening;
* Absence of a recent clinically-relevant progression of micro- and macro-vascular complications (see exclusion criteria);
* Written informed consent to participate to the study.

Exclusion criteria:

* Age below 35 years
* Type 1 diabetes or other causes of diabetes (pancreatectomy, gestational diabetes, etc.)
* HbA1c < 7% or ≥ 9% at the screening visit
* Treatment with any blood glucose lowering treatment other than Metformin in the six months before screening visit
* BMI < 20 or ≥ 40 kg/m2, or current/ past history of clinically-relevant eating disorders (including -but no limited to- nervous anorexia, bulimia, binge-eating disorders, etc.)
* Significant progression of diabetic macro-angiopathy or cardiovascular disease in the six months prior to study visit
* Significant progression of diabetic micro-angiopathy in the six months prior to study visit
* Organ failure or other severe diseases limiting life expectancy;
* Beginning, in the three months before screening visit, of any kind of drug which can modify glycemic levels (beta-blockers, diuretics…), or acute disease (acute infection, urinary tract infection…) in three months before screening visit
* History of inflammatory/infective/autoimmune chronic disease
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, gastric surgery, inflammatory bowel disease;
* Any clinically significant abnormality identified on physical examination, laboratory tests, ECG or vital signs at screening that in the judgment of the investigator would preclude safe completion of the study;
* Uncontrolled or inadequately controlled hypertension at screening (Systolic Blood Pressure (SBP)>190 or Diastolic Blood Pressure (DBP) >100 mmHg)
* Ongoing pregnancy or absence of effective contraception in women with childbearing potential
* Contraindications to the maintenance of the background therapy (Metformin), including -but not limited to- chronic kidney failure or plasma creatinine concentrations > 1.5 mg/dL, severe respiratory failure, etc.;
* Contraindications to the use of a Sulfonylurea;
* Contraindications to the use of a DPP-IV Inhibitor;
* Laboratory findings, or other disease conditions, at the screening visit that might interfere with study measurements:

  1. Hemoglobinopathy known to affect HbA1c assays;
  2. Known chronic liver diseases, including HBV (hepatitis B virus) and HCV (hepatitis C virus) infection;
  3. Liver makers (aspartate transaminase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), Gamma-glutamyltransferase (GGT) , bilirubin) above 2 times the upper normal limit;
  4. Amylase and/or lipase above 2 times the upper normal limit;
* Chronic use of systemic and/or inhaled corticosteroids (only topical corticosteroids are allowed);
* History of low compliance, clinically-relevant psychiatric disorders or any current/ historical finding suggesting the patient as inappropriate to follow the study procedures.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Zavaroni, MD, Principal Investigator — Azienda Ospedaliera-Universitaria di Parma
Locations (2):
- Italy (2):
  - Azienda Opedaliera-Universitaria, Parma
  - Azienda Ospedaliera-Universitaria, Parma

REFERENCES:
- [Derived] Dei Cas A, Spigoni V, Cito M, Aldigeri R, Ridolfi V, Marchesi E, Marina M, Derlindati E, Aloe R, Bonadonna RC, Zavaroni I. Vildagliptin, but not glibenclamide, increases circulating endothelial progenitor cell number: a 12-month randomized controlled trial in patients with type 2 diabetes. Cardiovasc Diabetol. 2017 Feb 23;16(1):27. doi: 10.1186/s12933-017-0503-0. PMID 28231835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals with type 2 diabetes were recruited in the outpatient Diabetes Unit of Parma University Hospital
Period: Overall Study
Arm/Group | Vildagliptin & Metformin | Glibenclamide & Metformin
Started | 40 (Received allocated intervention n=38 Did not receive allocated intervention (only metformin) n=2) | 24
Discontinued Intervention | 0 | 5
Completed | 40 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vildagliptin & Metformin | Glibenclamide & Metformin | Total
Number analyzed (Participants) | 40 | 24 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (9) | 63 (10) | 62 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 26 | 17 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 24 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 40 | 24 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 40 | 24 | 64
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 29.1 [26.8 to 32.9] | 28.9 [25.4 to 34.1] | 29.0 [26.2 to 33.9]
HBA1C [Median (Inter-Quartile Range); unit: %] | 7.7 [7.4 to 7.9] | 7.7 [7.5 to 8.1] | 7.7 [7.4 to 8.1]
Endothelial Progenitor Cells Number [Median (Inter-Quartile Range); unit: EPC/10^6 cells] | 39 [24.0 to 58.2] | 37.5 [25.0 to 59.8] | 38 [24.2 to 58.2]

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in the Endothelial Progenitor Cell (EPC) Number
Description: The study primary endpoint was the change from baseline values of the EPC number in the Vildagliptin vs Glibenclamide arm at 4 and 12 months.
Time Frame: V0, V2 (month 4), V4 (12 month)
Population: Intention to treat (ITT) analysis
Measure: Median (Inter-Quartile Range); unit: EPC/10^6 cells
Arm/Group | Vildagliptin & Metformin | Glibenclamide & Metformin
Number analyzed (Participants) | 40 | 24
EPC/10^6 cells
  V2 (4 month) | 37 [27.0 to 65.0] | 36 [23.0 to 54.2]
  V4 (12 month) | 45 [29.7 to 67] | 32 [22.2 to 53.5]
Statistical Analysis 1: Comparison: Vildagliptin & Metformin vs Glibenclamide & Metformin; Test type: Other; p < 0.05, Regression, Linear; Generalized linear model (GLM)
Statistical Analysis 2: Comparison: Vildagliptin & Metformin vs Glibenclamide & Metformin; Test type: Superiority; p < 0.05, ANOVA; adjustment for baseline value of EPC; Slope = 0.362, 95% CI 2-sided [0.028 to 0.695]

2. Secondary Outcome: Absolute Change in HbA1C Compared to Baseline
Description: The secondary endpoint was the change from baseline values of HbA1C in the Vildagliptin vs Glibenclamide arm at 4 and 12 months
Time Frame: V0 (randomization), V2 (month4), V4 (month 12).
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Vildagliptin & Metformin | Glibenclamide & Metformin
Number analyzed (Participants) | 40 | 24
percentage
  V2 (4 month) | 6.8 [6.4 to 7.3] | 6.8 [6.4 to 7.3]
  V4 (12 month) | 7.0 [6.5 to 7.3] | 7.1 [6.5 to 7.5]
Statistical Analysis 1: Comparison: Vildagliptin & Metformin vs Glibenclamide & Metformin; Test type: Superiority; p < 0.05, ANOVA; Slope = -0.067, 95% CI 2-sided [-0.358 to 0.224]

ADVERSE EVENTS:
Time Frame: 4 months
Description: Hypoglycemia
Arm/Group | Vildagliptin & Metformin | Glibenclamide & Metformin
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/24
Other Adverse Events (participants affected / at risk) | 0/40 | 5/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vildagliptin & Metformin (N=40) | Glibenclamide & Metformin (N=24)
hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) — At each study visit side effects were systematically investigated and patients were asked to contact the centre in case of adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes